CLINICAL TRIAL: NCT04673669
Title: Validation of the Measurement of the Strength of the Posterior Tibial Muscle by Hand-held Dynamometer Against a Reference Isokinetic Dynamometer
Brief Title: Measurement of the Strength of the Posterior Tibial Muscle by Hand-held Dynamometer
Acronym: TPHHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020_60; 2020-A02675-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Valgus Foot Deformity
Keywords: Posterior tibial; hand-held dynamometer, isokinetics; isokinetics, measurement validation
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): measuring the strength of the tendon of the posterior tibial muscle in healthy subjects with a hand-held dynamometer by two examiners and with an isometric dynamometer
  Interventions: Diagnostic Test: Posterior tibial tendon strength mesure

INTERVENTIONS:
Diagnostic Test: Posterior tibial tendon strength mesure — Posterior tibial tendon strength is assessed with a hand-held dynamometer by two independent observer and with an isometric dynamometer by one observer.

SUMMARY:
Adult flat foot valgus is a degenerative pathology that causes damage to the ligaments of the hindfoot as well as dysfunction of the tendon of the posterior tibial muscle.

Currently, there is a lack of a tool allowing a standardized, reliable, reproducible and validated measurement of the strength of the tendon of the posterior tibial muscle in consultation of foot surgery.

The hand-held dynamometer could be that tool. The study would consist in measuring the strength of the tendon of the posterior tibial muscle in healthy subjects with a hand-held dynamometer (MicroFET2) by two examiners and compared to isometric reference measurements (CON-TREX CMV Multi-Joint) to validate the reliability of the measurement and its reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Patients from physical medicine and rehabilitation department hospitalized for pathologies other than neurological or osteo-articular pathologies affecting the lower limbs,
* Having no neurological or osteo-articular pathology affecting the lower limbs f one year,
* No history of surgery on the rear foot and ankle,
* Written informed consent from person,
* Socially insured patient person,
* Person willing to comply with all study procedures and study duration.

Exclusion Criteria:

* Neurological or osteo-articular pathologies affecting the lower limbs,
* Known pathologies of the tendon of the posterior tibialis muscle,
* Deformations of the foot (flat foot, hollow foot),
* History of hindfoot or ankle surgery,
* Pregnant or breastfeeding woman,
* Inability to receive information, consent and participate in the whole study,
* Person under judicial protection or deprived of liberty,
* Person participating in another clinical trial,
* No social insurance cover,
* No written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient of the inversion force (or supination measured in Newton) of the foot between the measurement made with the hand dynamometer and the measurement made with the isokinetic dynamometer (gold standard). | on the day of first evaluation (at day 1)
  Validity of the measurement of the tendon strength of the posterior tibial muscle with a hand-held dynamometer (MicroFET2) compared to the gold standard (CON-TREX CMV Multi-Joint) in subjects.

SECONDARY OUTCOMES:
Intra-class correlation coefficient of the inversion force of the foot between two measurements made by the same observer with the hand dynamometer (intra-observer reproducibility). | on the day of first evaluation (At day 1) and on the day of second evaluation (at day 2)
  the inversion force (or supination measured in Newton). The two measurements will be performed during two consultations one day apart.
Intra-class correlation coefficient of the inversion force of the foot between measurements made by two different observers with the hand dynamometer (intra-observer reproducibility). | on the day of first evaluation (At day 1) and on the day of second evaluation (at day 2)
  the inversion force (or supination measured in Newton)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Amouyel, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Salengro - Hopital B Chr Lille - Lille, Lille, France